CLINICAL TRIAL: NCT04389957
Title: Improving Colonoscopy Quality for Colorectal Cancer Screening in the National VA Healthcare System
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: SDR 18-148
Record Dates: First submitted 2020-05-06; First posted 2020-05-15 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Neoplasms
Keywords: Quality Improvement; Adenoma; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Endoscopy Providers: In the primary analysis model, there were 68 sites with usable data with 98,442 procedures from 445 providers in the pre-intervention time frame and 129,972 procedures from 392 providers in the post-intervention time frame.
  Interventions: Other: Veterans Affairs Endoscopy Quality Improvement Program (VA-EQuIP)

INTERVENTIONS:
Other: Veterans Affairs Endoscopy Quality Improvement Program (VA-EQuIP) — We created an innovative informatics framework for centralized reporting of colonoscopy quality across the VA, facilitating the implementation of the VA Endoscopy Quality Improvement Program (VA-EQuIP). The VA-EQuIP quality dashboard (updated at 6 month intervals) provided adenoma detection rates (ADR), bowel preparation quality, and cecal intubation rate to every facility.This initiative directly addressed the OIG's recommendations and the VA's urgent need for evidence-based colonoscopy quality measurement and reporting. Through VA-EQuIP, we provided bi-annual audits and feedback on colonoscopy quality for VA sites and endoscopists, along with individual provider benchmarking against local and national performance standards. Additionally, we organized collaborative learning sessions led by national experts in colonoscopy training and quality. These sessions focused on shared learning, featuring lectures, discussions, skill-building activities, and work on quality improvement projects.

SUMMARY:
High quality screening colonoscopy is critical for colorectal cancer (CRC) prevention in Veterans. There is significant variability in colonoscopy quality in VA that is directly linked to differences in CRC incidence and death. The investigators developed the VA Endoscopy Quality Improvement Program (VA-EQuIP) that the National GI program office will implement using centralized quality measurement and reporting for adenoma detection rates (ADR), bi-annual audit and feedback with provider benchmarking to local and national performance, and collaborative learning to support colonoscopy quality improvement. Using a cluster randomized controlled trial, the investigators will study the implementation of VA-EQuIP and determine the efficacy of its intervention on adenoma detection rates, which are directly linked to CRC incidence and death.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) prevention is a top VA priority. Veterans are highly impacted by CRC, the third most common cancer diagnosed with a 3-year mortality rate of 35%. Colonoscopy screening can save lives, and is the cornerstone of effective prevention. The National Polyp Study showed that removal of adenomas during screening colonoscopy decreases the subsequent development of CRC by up to 90% and death by up to 50% in comparison to historical controls. In VA, colonoscopy is the primary CRC screening modality with over 200,000 colonoscopies performed each year. Eighty-two percent of Veterans are up-to-date on CRC screening, with 89% having a colonoscopy. However, the quality of those VA colonoscopies is unknown.

High quality colonoscopy is critical for CRC prevention. Observational studies found significant rates of CRC even after normal colonoscopy, likely due to colonoscopists' varied performance in detecting and removing polyps. Among Medicare beneficiaries, approximately 7% of all CRC occurred in individuals who had colonoscopy that apparently missed the CRC diagnosis. A pooled analysis from eight surveillance studies suggested 52% of incident CRCs after colonoscopy were due to missed lesions. These interval cancers highlight the need to focus on colonoscopy quality indicators.

Adenoma detection rate (ADR) significantly varies by provider and has been strongly linked to both CRC incidence and mortality. In essence, polyps that are not found cannot be removed for CRC prevention. ADR, defined as the proportion of screening colonoscopies performed by a physician that has one or more histologically-confirmed adenomatous polyps or CRC, is the primary benchmark for colonoscopy inspection quality. Increasing ADR correlates with a lower risk of interval and fatal CRC. A landmark US study of 314,872 colonoscopy exams showed marked variability in providers' ability to detect polyps, with the ADR ranging from 7.4 to 52.5%. In patients of providers with the highest ADRs, as compared with those in the lowest, the adjusted hazard ratios (HR) for fatal interval CRC was 0.38 (95% Confidence Interval [CI], 0.22 to 0.65). Each 1% increase in ADR was associated with a decrease risk of 3% for interval CRC and 5% for CRC death.

Using the methods the team developed, the investigators have powerful pilot results showing colonoscopy quality variability in the VA and direct association with CRC death. From 1999-2011, there were 634,331 Veterans with baseline colonoscopy performed by one of 3101 colonoscopists with ADRs ranging from 13-79%. In patients who had a colonoscopy without polyps found, the higher the provider ADR, the more protected the patient was from developing future CRC: adjusted HR (adjHR) 0.57 for incident (95%CI: 0.42-0.79; ptrend< 0.001) and 0.73 for fatal (95%CI: 0.50-1.06; p=0.047) CRC for the highest vs. lowest ADR quintile. Among individuals who had a colonoscopy with polypectomy, increasing ADR was also associated with reduced risk: adjHRs 0.46 for incident (95%CI: 0.34-0.62; ptrend< 0.001) and 0.53 for fatal (95%CI: 0.34-0.84; ptrend=0.006) CRC for the highest vs. lowest quintile. A 5% absolute increase in ADR was associated with relative reductions in fatal CRC risk of 4% after normal colonoscopy (adjHR 0.96, 95%CI: 0.95-0.97) and 6% after polypectomy (adjHR 0.94; 95%CI: 0.89-0.98) Other important quality metrics, including bowel preparation quality and cecal intubation rate also impact patient outcomes with poor bowel preparation and incomplete examinations associated with missed lesions and need for earlier repeat procedures.

Audit and feedback of colonoscopy quality improves performance and outcomes. The VA Surgical Quality Improvement Program (VASQIP) is an example of a VA nationwide reporting system that formed to focus on quality and has led to a decrease in mortality of 47% in patients 30 days after surgery. VASQIP provides information to providers for self-assessment and quality improvement purposes. There is similarly strong evidence that providing colonoscopy performance feedback improves quality and patient outcomes. Kahi and colleagues showed in a single-center VA setting that a quarterly report card improved colonoscopy quality. Most recently, in a large prospective European cohort study evaluating annual feedback and quality benchmark indicators on screening colonoscopy performance, the majority of the endoscopists (74.5%) increased their annual ADR. Moreover, individuals examined by endoscopists in the highest ADR quintile (> 24.6%) had significantly lower risk of interval CRC and death. When compared with no increase in ADR, reaching or maintaining the highest quintile ADR decreased adjusted hazard ratios for interval and fatal CRC to 0.27 (95% CI, 0.12-0.63; p = .03), and 0.18 (95% CI, 0.06-0.56; p = .03).

Quality Gap: Quality reporting improves patient outcomes. The national VA healthcare system currently lacks a reliable, efficient program to routinely measure and report colonoscopy quality. Accurate measurement of quality metrics is challenging, because validated quality metrics are not available in structured VA data from VA Corporate Data Warehouse (CDW). The challenge is multifactorial. Colonoscopy procedure documentation resides in text notes in Vista/ Computerized Patient Record System (CPRS) or endoscopic reporting software. The commonly used VA endoscopy note writer software programs (i.e. Endopro®, Provation®, etc) do not facilitate tracking pathology data and quality measurement. None of the current VA endoscopy reporting programs link to VA pathology data (to determine ADR); and production-level pathology data is not in the CDW. Thus, within VA, there has not been a reliable, efficient way to track critical procedure and pathology results to measure colonoscopy quality and ensure optimal protection from CRC incidence and death for Veterans.

Proposed Solution and Rationale for Study: The foundation of VA-EQuIP is a novel natural language processing (NLP) algorithm and informatics reporting infrastructure that the investigators developed to measure the quality of colonoscopies performed by individual VA colonoscopists. The team will evaluate a national quality improvement program to better understand how and why such a program is effective or ineffective in different contexts. This study is critically needed to allow us to perform a rigorous evaluation to answer implementation science questions and to advance the clinical and epidemiologic knowledge on the impact of colonoscopy quality on CRC mortality. Leveraging the informatics investment made by VA Health Services Research and Development Service (HSR&D) as well as the National Gastroenterology Program office partnership in quality improvement initiatives, the roll out of VA-EQuIP is a rare opportunity to study, in real time, the deployment and impact of a large-scale learning health system initiative. Most existing performance measures are calculated at the facility level. The concept of calculating metrics from individual provider procedures and comparing these metrics not only with local peers but with national providers represents a profound culture shift. This is where implementation science becomes essential, especially with respect to stakeholder engagement, adaptation and tailoring.

A primary justification for this study is that VA-EQuIP has a high probability of improving a quality metric outcome (ADR) directly associated with CRC death, one of the most common cancers in Veterans. A randomized controlled trial of this magnitude is an opportunity to show, for the first time, that even small improvements in clinical performance from audit and feedback can save Veterans lives, since even a 1% increase in ADR translates to a 3% reduction in interval cancer death. The proposal for a randomized program evaluation is a tremendous opportunity to determine the large scale effect of the audit and feedback strategy on changes in the colonoscopy quality metrics of individual endoscopists over time. The evaluation of VA-EQuIP implementation will identify factors associated with effective implementation and colonoscopy quality improvement (impact) at VA sites. Prior and planned work builds toward long-term goal to reduce mortality in Veterans by increasing early detection of CRC and inform national quality improvement initiatives such as remediation training for continual low performing endoscopists.

Finally, with upcoming expansion to community care, VA will be making policy decisions about what services should be furnished by VA versus non-VA providers. It is more crucial than ever that health services researchers apply rigorous methods to identify meaningful quality metrics that are linked by evidence to patient outcomes so that these measures of quality will be used to justify such crucial "make versus buy" determinations. It is hopeful that the investigators study will not only improve colonoscopy quality but also provide a framework for assessing the quality of other procedures such as bone marrow biopsy or bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Quantitative surveys will be delivered to endoscopy or GI section chiefs responsible for endoscopy services for each enrolled site.
* Qualitative interviews will be conducted with GI section chiefs and individual endoscopists at participating facilities.
* A list of criteria for selection of participants in the clinical study, provided in terms of inclusion and exclusion criteria is suitable for assisting potential participants in identifying clinical studies of interest.
* All VA facilities with existing colonoscopy procedure or pathology notes in our operational database.

Exclusion Criteria:

-VA facilities without existing colonoscopy procedure or pathology notes in our operational database will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Researchers will recruit section chiefs and endoscopists at eligible sites. Colonoscopy quality data will be delivered to providers and GI section chiefs. Surveys and interviews will be delivered to identified local endoscopists and GI section chiefs responsible for endoscopy services potentially eligible VA sites.
Sampling Method: Non-Probability Sample
Enrollment: 445 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Gawron, MD MS, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT; Tonya R. Kaltenbach, MD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (6):
- United States (6):
  - VA San Diego Health Care System, San Diego, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - Richard L. Roudebush VA Medical Center, Indianapolis, Indiana
  - VA Ann Arbor Health Care System, Ann Arbor, Michigan
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - VA Puget Sound Health Care System, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gawron AJ, Yao Y, Gupta S, Cole G, Whooley MA, Dominitz JA, Kaltenbach T. Simplifying Measurement of Adenoma Detection Rates for Colonoscopy. Dig Dis Sci. 2021 Sep;66(9):3149-3155. doi: 10.1007/s10620-020-06627-2. Epub 2020 Oct 8. PMID 33029706
- [Background] Gawron AJ, Sultan S, Glorioso TJ, Califano S, Kralovic SM, Jones M, Kirsh S, Dominitz JA. Pre-endoscopy coronavirus disease 2019 screening and severe acute respiratory syndrome coronavirus-2 nucleic acid amplification testing in the Veterans Affairs healthcare system: clinical practice patterns, outcomes, and relationship to procedure volume. Gastrointest Endosc. 2022 Sep;96(3):423-432.e7. doi: 10.1016/j.gie.2022.04.018. Epub 2022 Apr 22. PMID 35461889
- [Background] Gawron AJ, Dominitz JA. Higher Quality Colonoscopy: Worth the Wait? Clin Transl Gastroenterol. 2022 Apr 1;13(4):e00471. doi: 10.14309/ctg.0000000000000471. PMID 35297791
- [Background] Gupta S, Earles A, Bustamante R, Patterson OV, Gawron AJ, Kaltenbach TR, Yassin H, Lamm M, Shah SC, Saini SD, Fisher DA, Martinez ME, Messer K, Demb J, Liu L. Adenoma Detection Rate and Clinical Characteristics Influence Advanced Neoplasia Risk After Colorectal Polypectomy. Clin Gastroenterol Hepatol. 2023 Jul;21(7):1924-1936.e9. doi: 10.1016/j.cgh.2022.10.003. Epub 2022 Oct 19. PMID 36270618
- [Background] Demb J, Liu L, Bustamante R, Dominitz JA, Earles A, Shah SC, Gawron AJ, Martinez ME, Gupta S. COVID-19 Pandemic Had Minimal Impact on Colonoscopy Completion After Colorectal Cancer Red Flag Sign or Symptoms in US Veterans. Dig Dis Sci. 2023 Apr;68(4):1208-1217. doi: 10.1007/s10620-022-07685-4. Epub 2022 Sep 28. PMID 36169748
- [Background] Gawron AJ, Bailey T, Codden R, Dominitz J, Gupta S, Helfrich C, Kahi C, Krop L, Malvar C, McKee G, Millar M, Mog A, Nguyen-Vu T, Patterson O, Presson AP, Saini S, Whooley M, Yao Y, Zickmund S, Kaltenbach T. Improving colonoscopy quality in the national VA healthcare system. Contemp Clin Trials. 2025 Feb;149:107784. doi: 10.1016/j.cct.2024.107784. Epub 2024 Dec 25. PMID 39730079
- [Background] Gawron AJ, Mckee G, Dominitz JA, Yao Y, Whooley M, Kaltenbach T. Validation of a National Pathology Database for Colonoscopy Quality Reporting and Assurance. Clin Gastroenterol Hepatol. 2025 Apr;23(5):866-868.e1. doi: 10.1016/j.cgh.2024.08.017. Epub 2024 Aug 28. No abstract available. PMID 39209190
- [Background] Kaltenbach T, Gawron A, Meyer CS, Gupta S, Shergill A, Dominitz JA, Soetikno RM, Nguyen-Vu T, A Whooley M, Kahi CJ. Adenoma Detection Rate (ADR) Irrespective of Indication Is Comparable to Screening ADR: Implications for Quality Monitoring. Clin Gastroenterol Hepatol. 2021 Sep;19(9):1883-1889.e1. doi: 10.1016/j.cgh.2021.02.028. Epub 2021 Feb 19. PMID 33618027
- [Background] Trivedi M, Godil S, Demb J, Earles A, Bustamante R, Patterson OV, Gawron AJ, Kaltenbach T, Mahata S, Liu L, Gupta S. Baseline Characteristics and Longitudinal Outcomes of Traditional Serrated Adenomas: A Cohort Study. Clin Gastroenterol Hepatol. 2023 Jun;21(6):1637-1645. doi: 10.1016/j.cgh.2022.09.030. Epub 2022 Oct 12. PMID 36243354
- [Background] Gawron AJ, Horner B, Zurbuchen R, Boynton K, Fang JC. A comprehensive intervention to enhance inpatient colon preparation quality for colonoscopy. Minerva Gastroenterol (Torino). 2023 Sep;69(3):351-358. doi: 10.23736/S2724-5985.21.02766-5. Epub 2021 Apr 1. PMID 33793164

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sites could be included in the study if we could identify colonoscopy procedure and pathology notes in the VA central data warehouse (CDW) database for providers at the site. Of the 151 VA sites, there were 68 sites with reliable colonoscopy and pathology data from the CDW with 98,442 procedures from 445 providers. In the post-intervention time frame, we collected data from 129,972 procedures and 392 providers.
Units Other Than Participants: VA-EQuIP Sites
Groups:
- Wedge 1 - 6 Months Baseline, 24 Months VA-EQuIP: Wedge 1 included 14 sites and 84 providers. Our intervention effect was estimated with the pre-intervention timepoint defined as 1/1/21 through dashboard release at the site. The intervention began at dashboard release and concluded in 6/30/23. The post-intervention timepoint was defined as beginning 3 months post dashboard release to 6/30/23.
- Wedge 2 - 9 Months Baseline, 21 Months VA-EQuIP: Wedge 2 included 14 sites and 83 providers. Our intervention effect was estimated with the pre-intervention timepoint defined as 1/1/21 through dashboard release at the site. The intervention began at dashboard release and concluded in 6/30/23. The post-intervention timepoint was defined as beginning 3 months post dashboard release to 6/30/23.
- Wedge 3 - 12 Months Baseline, 18 Months VA-EQuIP: Wedge 3 included 14 sites and 93 providers. Our intervention effect was estimated with the pre-intervention timepoint defined as 1/1/21 through dashboard release at the site. The intervention began at dashboard release and concluded in 6/30/23. The post-intervention timepoint was defined as beginning 3 months post dashboard release to 6/30/23.
- Wedge 4 - 15 Months Baseline, 15 Months VA-EQuIP: Wedge 4 included 13 sites and 97 providers. Our intervention effect was estimated with the pre-intervention timepoint defined as 1/1/21 through dashboard release at the site. The intervention began at dashboard release and concluded in 6/30/23. The post-intervention timepoint was defined as beginning 3 months post dashboard release to 6/30/23.
- Wedge 5 - 18 Months Baseline, 12 Months VA-EQuIP: Wedge 5 included 13 sites and 88 providers. Our intervention effect was estimated with the pre-intervention timepoint defined as 1/1/21 through dashboard release at the site. The intervention began at dashboard release and concluded in 6/30/23. The post-intervention timepoint was defined as beginning 3 months post dashboard release to 6/30/23.
Period: Overall Study
Arm/Group | Wedge 1 - 6 Months Baseline, 24 Months VA-EQuIP | Wedge 2 - 9 Months Baseline, 21 Months VA-EQuIP | Wedge 3 - 12 Months Baseline, 18 Months VA-EQuIP | Wedge 4 - 15 Months Baseline, 15 Months VA-EQuIP | Wedge 5 - 18 Months Baseline, 12 Months VA-EQuIP
Started | 84; 14 VA-EQuIP Sites | 83; 14 VA-EQuIP Sites | 93; 14 VA-EQuIP Sites | 97; 13 VA-EQuIP Sites | 88; 13 VA-EQuIP Sites
Completed | 77; 14 VA-EQuIP Sites | 76; 14 VA-EQuIP Sites | 81; 14 VA-EQuIP Sites | 77; 13 VA-EQuIP Sites | 81; 13 VA-EQuIP Sites
Not Completed | 7; 0 VA-EQuIP Sites | 7; 0 VA-EQuIP Sites | 12; 0 VA-EQuIP Sites | 20; 0 VA-EQuIP Sites | 7; 0 VA-EQuIP Sites
Not completed — Providers without data in the post intervention timeframe. | 7 | 7 | 12 | 20 | 7

BASELINE CHARACTERISTICS:
Population: For the 68 included sites, there were 98,442 colonoscopy procedures from 445 providers in the pre-intervention time frame.
Groups:
- Providers: In the primary analysis model, there were 68 sites with usable data with 98,442 procedures from 445 providers in the pre-intervention time frame and 129,972 procedures from 392 providers in the post-intervention time frame.
Arm/Group | Providers
Number analyzed (Participants) | 445
Age, Customized [Count of Participants; unit: Participants] — Population: Information about age was unavailable for 5 providers.
  Participants
    Age Groups: number analyzed (Participants) | 440
    Age Groups: 39 years or younger | 97
    Age Groups: 40-49 years | 129
    Age Groups: 50-59 years | 94
    Age Groups: 60 years or older | 120
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Information about sex was unavailable for 6 providers
  Participants
    number analyzed (Participants) | 439
    Female | 116
    Male | 323
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Continental | 40
  United States: Midwest | 136
  United States: North Atlantic | 99
  United States: Pacific | 103
  United States: Southeast | 67
Specialty [Count of Participants; unit: Participants]
  Gastroenterology | 390
  Surgery | 55
Years since completion of medical degree [Count of Participants; unit: Participants] — Population: Information about completion of medical degree was unavailable for 27 providers.
  Participants
    number analyzed (Participants) | 418
    Less than 10 years | 49
    10-19 years | 128
    20-29 years | 99
    30-39 years | 83
    40 or more years | 59

OUTCOME MEASURES:

1. Primary Outcome: Provider Adenoma Detection Rate (for All Colonoscopies)
Description: Adenoma detection rate is a provider level quality metric. For individual endoscopy providers, the numerator is the number of patients undergoing colonoscopy for any indication in which one or more adenomatous polyps were removed. The denominator is the total number of patients undergoing colonoscopy for each individual provider. Data will be obtained from our operational database for quality measurement and reporting.
Time Frame: Our intervention effect was estimated with the pre-intervention timepoint defined as 1/1/21 through dashboard release at the site, and post-intervention timepoint defined as beginning 3 months post dashboard release and concluding 6/30/23.
Population: We assessed the adenoma detection rate of 445 providers in the pre-intervention time frame and 392 providers in the post-intervention time frame.
Measure: Mean (Standard Deviation); unit: % of colonoscopies w/ 1+ adenomas
Units Other Than Participants: VA-EQuIP Sites
Groups:
- Wedge 1: Wedge 1 included 14 sites and 84 providers in the pre-intervention time frame and 14 sites and 77 providers in the post-intervention time frame.
- Wedge 2: Wedge 2 included 14 sites and 83 providers in the pre-intervention time frame and 14 sites and 76 providers in the post-intervention time frame.
- Wedge 3: Wedge 3 included 14 sites and 93 providers in the pre-intervention time frame and 14 sites and 81 providers in the post-intervention time frame.
- Wedge 4: Wedge 4 included 13 sites and 97 providers in the pre-intervention time frame and 13 sites and 77 providers in the post-intervention time frame.
- Wedge 5: Wedge 5 included 13 sites and 88 providers in the pre-intervention time frame and 13 sites and 81 providers in the post-intervention time frame.
Arm/Group | Wedge 1 | Wedge 2 | Wedge 3 | Wedge 4 | Wedge 5
Number analyzed (Participants) | 84 | 83 | 93 | 97 | 88
Number analyzed (VA-EQuIP Sites) | 14 | 14 | 14 | 13 | 13
% of colonoscopies w/ 1+ adenomas
  Pre-Intervention | 52.7 (13.7) | 46.9 (12.4) | 43.5 (15.0) | 42.8 (18.2) | 45.6 (12.3)
  Post-Intervention: number analyzed (Participants) | 77 | 76 | 81 | 77 | 81
  Post-Intervention | 50.9 (16.7) | 52.0 (12.6) | 46.2 (11.2) | 49.5 (14.3) | 50.9 (12.6)

2. Secondary Outcome: Bowel Preparation Quality (Provider Level)
Description: Bowel preparation quality is determined by each endoscopist for bowel cleanliness allowing polyp visualization and removal. Bowel preparation quality is measured as Adequate or Inadequate by our quality reporting system. For each provider, bowel preparation quality will be calculated with the numerator equal to all colonoscopies with "adequate" preparation quality divided by the denominator of all colonoscopies performed by the provider.
Time Frame: as for outcome 1
Population: We assessed bowel preparation quality of 445 providers in the pre-intervention time frame and 392 providers in the post-intervention time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Wedge 1 | Wedge 2 | Wedge 3 | Wedge 4 | Wedge 5
Number analyzed (Participants) | 84 | 83 | 93 | 97 | 88
Participants
  Pre-Intervention: Less than 85% | 19 | 21 | 48 | 50 | 44
  Pre-Intervention: 85% or greater | 65 | 62 | 45 | 47 | 44
  Post-Intervention: number analyzed (Participants) | 77 | 76 | 81 | 77 | 81
  Post-Intervention: Less than 85% | 20 | 16 | 36 | 47 | 28
  Post-Intervention: 85% or greater | 57 | 60 | 45 | 30 | 53

3. Secondary Outcome: Cecal Intubation Rate (Provider Level) - Revision
Description: Cecal intubation is a provider level quality metric. The cecal intubation rate is the proportion of colonoscopies with cecal intubation documented in the procedure note.
Time Frame: as for outcome 1
Population: We assessed cecal intubation rate of 445 providers in the pre-intervention time frame and 392 providers for the post-intervention time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Wedge 1 | Wedge 2 | Wedge 3 | Wedge 4 | Wedge 5
Number analyzed (Participants) | 84 | 83 | 93 | 97 | 88
Participants
  Pre-Intervention: Less than 90% | 16 | 22 | 41 | 51 | 31
  Pre-Intervention: 90% and greater | 68 | 61 | 52 | 46 | 57
  Post-Intervention: number analyzed (Participants) | 77 | 76 | 81 | 77 | 81
  Post-Intervention: Less than 90% | 17 | 7 | 32 | 31 | 36
  Post-Intervention: 90% and greater | 60 | 69 | 49 | 46 | 45

ADVERSE EVENTS:
Time Frame: Data collection spans 30 months
Description: There were no serious risks of adverse events anticipated in association with participation in the study. The intervention is a quality improvement program designed to provide providers with the opportunity to review their colonoscopy quality data and engage in shared learning sessions.
Groups:
- Providers: For the 68 included sites in the stepped-wedge trial, we assessed 445 providers with 98,442 procedures in the pre-intervention time frame and 392 providers with 129,972 procedures in the post-intervention time frame.
Arm/Group | Providers
All-Cause Mortality (participants affected / at risk) | 0/445
Serious Adverse Events (participants affected / at risk) | 0/445
Other Adverse Events (participants affected / at risk) | 0/445

LIMITATIONS AND CAVEATS:
Limitations include inability to access data from every VA facility. The coronavirus disease (COVID-19) pandemic did result in a minor delay to the start of the trial but we were able to complete the trial on time and data analysis occurred with a no-cost extension.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT04389957/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT04389957/ICF_001.pdf